CLINICAL TRIAL: NCT00196885
Title: Effect of N-Acetylcysteine on Skeletal Muscle in Cachectic Cancer Patients Undergoing a Resistance Training Program (Phase 2 Study)
Brief Title: Effect of an Antioxidant on Cancer-Cachectic Patients Undergoing Exercise Training
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: whilde157/2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Gastrointestinal Neoplasms; Bronchial Carcinoma; Hodgkin Disease; Non-Hodgkin Lymphoma; Weight Loss
Keywords: cancer cachexia; muscle wasting; weight loss; proteolysis
MeSH Terms: conditions — Gastrointestinal Neoplasms; Carcinoma, Bronchogenic; Hodgkin Disease; Lymphoma, Non-Hodgkin; Weight Loss; Muscular Atrophy | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine

SUMMARY:
The purpose of the study is to tests the hypothesis, that N-acetylcysteine (a thiol-antioxidant)improves the exercise training effect on cancer patients that experience weight loss (cachexia) as assessed by muscle mass and function as well as histomorphology.

ELIGIBILITY:
Inclusion Criteria:

* gastrointestinal or bronchial cancer
* weight loss of 10% within 6 months
* sufficient mobility

Exclusion Criteria:

* severe pain, steroid therapy, severe internal, muscular, neurological, psychiatric disease, N-acetylcysteine allergy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
muscle cross-sectional area, peak forces

SECONDARY OUTCOMES:
muscle fiber composition (biopsy vastus lateralis muscle mRNA levels of cytokines, myostatin. Activity of Akt-dependent pathways
muscle 31Phospho-magnetic-resonance spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Wulf Hildebrandt, MD, Study Director — German Cancer Research Center
Locations (1):
- German Cancer Research Center, D020, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Hauer K, Hildebrandt W, Sehl Y, Edler L, Oster P, Droge W. Improvement in muscular performance and decrease in tumor necrosis factor level in old age after antioxidant treatment. J Mol Med (Berl). 2003 Feb;81(2):118-25. doi: 10.1007/s00109-002-0406-7. Epub 2003 Feb 8. PMID 12601528